CLINICAL TRIAL: NCT03200223
Title: A Study of the Management of the Patient's Disease Based on the Life Log Data of Patient With Lifestyle-related Diseases Through a Wearable Device and Mobile App
Brief Title: Lifestyle Related Disease Management With Wearable Device and Mobile Application
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was completed
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Whun Kim, Clinical professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1706/405-301
Record Dates: First submitted 2017-06-25; First posted 2017-06-27 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Life Style Induced Illness
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized lifestyle intervention group (Experimental): Personalized lifestyle intervention group Patients who use mobile healthcare service application and receive personal feedback from clinician
  Interventions: Behavioral: Personalized healthcare service
- Conventional group (No Intervention): Patients with conventional care

INTERVENTIONS:
Behavioral: Personalized healthcare service — Personalized healthcare service, such as exercise recommendation, lifestyle activity coaching, health data monitoring
  Arms: Personalized lifestyle intervention group

SUMMARY:
In order to study the effectiveness of personalized healthcare intervention for lifestyle-related diseases, investigators designed this study using mobile application and clinical feedback coaching.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must agree to support by him/herself at enroll time
* Patient without severe cardiopulmonary disease, cancer, or other acute diseases
* Patient must be over BMI > 23 kg/m2

Exclusion Criteria:

* Patient who did not agree with this study
* Patient with severe cardiopulmonary disease, cancer, or other acute diseases
* Patient who are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Weight change | Baseline and after 2 weeks, 4 weeks of lifestyle modification
  Measuring weight change

SECONDARY OUTCOMES:
Body composition change | Baseline and after 2 weeks, 4 weeks of lifestyle modification
  Measuring body composition
Laboratory test result change | Baseline and after 2 weeks, 4 weeks of lifestyle modification
  Obstructive sleep apnea test

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Whun Kim, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JW, Ryu B, Cho S, Heo E, Kim Y, Lee J, Jung SY, Yoo S. Impact of Personal Health Records and Wearables on Health Outcomes and Patient Response: Three-Arm Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jan 4;7(1):e12070. doi: 10.2196/12070. PMID 30609978